CLINICAL TRIAL: NCT01406210
Title: Prospective and Retrospective Study to Develop a Multi-center Randomized Study, to Determine if Prevention of GERD Related Aspiration by Surgical Fundoplication Improves Lung Allograft Function
Brief Title: RESULT (REflux Surgery in Lung Transplantation) Preliminary Study Protocol
Acronym: RESULT
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00025618; 1R34HL105422-01 (NIH)
Record Dates: First submitted 2011-06-28; First posted 2011-08-01 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Reflux; Gastroesophageal Reflux Disease (GERD)
Keywords: Lung Transplant; REflux Surgery; Gastroesophageal Reflux Disease (GERD); Fundoplication
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples Without DNA — The bronchiolar lavage fluid (BALF) will be drawn during the bronchoscopy site and approximately up to 10 ml of the bronchiolar lavage (BAL) fluid will be placed in 7 storage vials (approximately 1.5 ml per vial), frozen using liquid nitrogen as the freezing agent, and shipped on dry ice to Duke University Medical Center and/or University of Toronto. Frozen samples will be stored at -80 °C to -85 °C until shipping, and the time between collection and freezing will be recorded.
  The tests used to assess the bronchiolar lavage fluid (BALF) may include, but are not limited to the following: Gastrin, Pepsinogen I, Pepsinogen II, Lipopolysaccharide (LPS), Bile acids (colorimetric and enzymatic approaches), and proteome assessment by mass spectrometry.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospective Group: Those patients that will be consented and data collected prospectively
- Retrospective Group: Those charts that will be utilized to collect retrospective data, waiver of consent will be granted by the IRBs.

SUMMARY:
The purpose of the prospective study is to collect information surrounding lung transplant in order to develop a randomized study to determine if prevention of gastroesophageal reflux disease (GERD) related aspiration (stomach acid coming up from the stomach into the esophagus) by surgical fundoplication improves lung rejection. Lung transplantation has evolved into an effective treatment for patients with end-stage lung disease; however, a significant limitation to long-term survival is patients develop a condition of scarring known as chronic lung rejection, which can cause lung function to deteriorate, thereby reducing a patient's chances for survival. Preliminary research has shown a correlation between the presence of gastroesophageal reflux disease (GERD) and impaired early lung rejection as assessed by a breathing test, FEV1 (the amount of forced expired air volume in 1 second).

The Investigator is interested in learning more about this condition and the potential for aspiration (inhaling fluid) injury. The primary goal of this preliminary study will be to identify aspiration markers that are correlated with adverse clinical outcomes (increased early rejection, decreased FEV1) that may be used as inclusion criteria for the future randomized trial.

The purpose of the retrospective study is to collect information surrounding lung transplant in order to develop a randomized study to determine if prevention of gastroesophageal reflux disease (GERD) related aspiration (stomach acid coming up from the stomach into the esophagus) by surgical fundoplication improves lung rejection.

The goal of this retrospective data collection is to review the following:

1. subject outcome event rates for subjects with and without gastroesophageal reflux disease (GERD) for survival, Bronchiolitis Obliterans Syndrome (BOS), acute rejection and Forced Expiratory Volume in the first second (FEV-1),
2. the estimated treatment effect of fundoplication on the above event rates,
3. a threshold effect for Bronchiolitis Obliterans Syndrome (BOS) and/or death are more likely to occur at higher or more proximal acid or non-acid contact times.

This data will be collected in order to better design and coordinate a multicenter prospective study.

DETAILED DESCRIPTION:
Prospective Group: Approximately 125 Bronchoalveolar Lavage (BAL) samples will be collected from eligible subjects at the time of clinical bronchoscopies and will be within 2 weeks of their esophageal study. The Bronchoalveolar Lavage (BAL) samples will be assayed for bile acids; pepsin, pepsinogen I and II; trypsin; gastrin, and Lipopolysaccharide (LPS) content. Short-term clinical outcome measures including acute rejection episodes, and Forced Expiratory Volume in the first second (FEV-1) at one year will be collected. Correlation between markers of reflux and aspiration will be analyzed.

Retrospective Group: Up to 800 charts within the past 5 years will be reviewed for 1) subject outcome event rates for subjects with and without Gastroesophageal Reflux Disease (GERD) for survival, Bronchiolitis Obliterans Syndrome (BOS), acute rejection and Forced Expiratory Volume in the first second (FEV-1), 2) what is the estimated treatment effect of fundoplication on the above event rates, 3) is there a threshold effect such that events such as BOS and death are more likely to occur only at higher or more proximal acid or non-acid contact times. This review will better address the role of Gastroesophageal Reflux Disease (GERD) in lung allograft failure, the clinical utility of surgical fundoplication in preventing lung allograft injury, and the role that acid and non-acid reflux as related to aspiration causes lung allograft injury as it relates to a wider population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female subject
2. 16 years of age
3. Recipient of a double-lung transplant
4. Previously have a 24-hour esophageal pH and/or impedance probe study within 12 months prior to transplant and/or within 12 months following transplantation. If the subject expired prior to 12 months from transplant date, they must have had a 24-hour esophageal pH and/or impedance probe study to be eligible in the study.

Exclusion Criteria:

1. Recipient of a single-lung transplant
2. Recipient of a re-do lung transplant
3. Recipient of a double-lung/heart or double-lung/ other organ transplant
4. Do not have a 24-hour esophageal pH and/or impedance probe study within 12 months pre-transplant or within 12 months following transplantation. The subject expired less than 12 months post transplant without having a 24-hour esophageal pH and/or impedance probe study
5. No Spirometry data is available for the subject
6. Subject who is participating in any other interventional clinical study
7. Unable to provide written informed consent or participate in long-term follow-up

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or non-pregnant female subject ≥16 years of age with a double-lung transplant who have undergone a 24-hour esophageal pH and/orimpedance probe study within 12 months prior to transplant and/or within 12 months following transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 647 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
BAL aspiration markers | 1 year
  For the prospective study analysis, we will be assessing the relationship of gastroesophageal reflux and aspiration post lung transplantation with the occurrence of lung allograft dysfunction by reviewing BAL samples prospectively collected in approximately 125 subjects. These BAL samples will be assayed for bile acids; pepsin, pepsinogen I and II; trypsin; gastrin, and LPS content. The correlation of the aspiration biomarkers to acute rejection, BOS, death and FEV-1 at one year will be assessed.
Death | 1 year
  For the retrospective study, the first specific goal of data collection is outcome event rates for subjects with and without GERD for survival and the estimated treatment effect of fundoplication on the above event rates. A threshold effect for death is more likely to occur at higher or more proximal acid or non-acid contact times. Up to 5 years of follow-up data will be available for analysis with the primary comparison at one year. These data will be used to better design and coordinate a multicenter prospective study.
BOS | 1 year
  For the retrospective study, the second specific goal of data collection is event rates for subjects with and without GERD for BOS and the estimated treatment effect of fundoplication on the above event rates. A threshold effect for BOS is more likely to occur at higher or more proximal acid or non-acid contact times. Up to 5 years of follow-up data will be available for analysis with the primary comparison at one year. These data will be used to better design and coordinate a multicenter prospective study.
FEV-1 | 1 year
  For the retrospective study, the third goal of data collection is evaluation of FEV-1 changes for subjects with and without GERD and the estimated treatment effect of fundoplication. Up to 5 years of follow-up data will be available for analysis with the primary comparison at one year. Data will be used to design a multicenter prospective study, address the role of GERD in lung allograft failure, the clinical utility of surgical fundoplication in preventing lung allograft injury, and the role that acid and non-acid reflux as related to aspiration causes lung allograft injury.
Acute Rejection | 1 year
  For the retrospective study, the final goal of data collection is evaluation of acute rejection episodes for subjects with and without GERD and the estimated treatment effect of fundoplication. Up to 5 years of follow-up data will be available for analysis with the primary comparison at one year. Data will be used to design a multicenter prospective study and to address the role of GERD in lung allograft failure, the clinical utility of surgical fundoplication in preventing lung allograft injury, and the role that acid and non-acid reflux as related to aspiration causes lung allograft injury.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Davis, MD, Principal Investigator — Duke University; Scott Palmer, MD, Principal Investigator — Duke University
Locations (4):
- United States (3):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Background] Estenne M, Maurer JR, Boehler A, Egan JJ, Frost A, Hertz M, Mallory GB, Snell GI, Yousem S. Bronchiolitis obliterans syndrome 2001: an update of the diagnostic criteria. J Heart Lung Transplant. 2002 Mar;21(3):297-310. doi: 10.1016/s1053-2498(02)00398-4. No abstract available. PMID 11897517
- [Background] Cooper JD, Billingham M, Egan T, Hertz MI, Higenbottam T, Lynch J, Mauer J, Paradis I, Patterson GA, Smith C, et al. A working formulation for the standardization of nomenclature and for clinical staging of chronic dysfunction in lung allografts. International Society for Heart and Lung Transplantation. J Heart Lung Transplant. 1993 Sep-Oct;12(5):713-6. PMID 8241207
- [Background] Kroshus TJ, Kshettry VR, Savik K, John R, Hertz MI, Bolman RM 3rd. Risk factors for the development of bronchiolitis obliterans syndrome after lung transplantation. J Thorac Cardiovasc Surg. 1997 Aug;114(2):195-202. doi: 10.1016/S0022-5223(97)70144-2. PMID 9270635
- [Background] Heng D, Sharples LD, McNeil K, Stewart S, Wreghitt T, Wallwork J. Bronchiolitis obliterans syndrome: incidence, natural history, prognosis, and risk factors. J Heart Lung Transplant. 1998 Dec;17(12):1255-63. PMID 9883768
- [Background] McKane BW, Trulock EP, Patterson GA, Mohanakumar T. Lung transplantation and bronchiolitis obliterans: an evolution in understanding. Immunol Res. 2001;24(2):177-90. doi: 10.1385/IR:24:2:177. PMID 11594455
- [Background] Boehler A, Estenne M. Obliterative bronchiolitis after lung transplantation. Curr Opin Pulm Med. 2000 Mar;6(2):133-9. doi: 10.1097/00063198-200003000-00009. PMID 10741773
- [Background] Snell GI, Esmore DS, Williams TJ. Cytolytic therapy for the bronchiolitis obliterans syndrome complicating lung transplantation. Chest. 1996 Apr;109(4):874-8. doi: 10.1378/chest.109.4.874. PMID 8635363
- [Background] Kesten S, Rajagopalan N, Maurer J. Cytolytic therapy for the treatment of bronchiolitis obliterans syndrome following lung transplantation. Transplantation. 1996 Feb 15;61(3):427-30. doi: 10.1097/00007890-199602150-00019. PMID 8610355
- [Background] Speich R, Boehler A, Russi EW, Weder W. A case report of a double-blind, randomized trial of inhaled steroids in a patient with lung transplant bronchiolitis obliterans. Respiration. 1997;64(5):375-80. doi: 10.1159/000196708. PMID 9311056
- [Background] Iacono AT, Keenan RJ, Duncan SR, Smaldone GC, Dauber JH, Paradis IL, Ohori NP, Grgurich WF, Burckart GJ, Zeevi A, Delgado E, O'Riordan TG, Zendarsky MM, Yousem SA, Griffith BP. Aerosolized cyclosporine in lung recipients with refractory chronic rejection. Am J Respir Crit Care Med. 1996 Apr;153(4 Pt 1):1451-5. doi: 10.1164/ajrccm.153.4.8616581.
- [Background] Dusmet M, Maurer J, Winton T, Kesten S. Methotrexate can halt the progression of bronchiolitis obliterans syndrome in lung transplant recipients. J Heart Lung Transplant. 1996 Sep;15(9):948-54. PMID 8889991
- [Background] Reichenspurner H, Meiser BM, Kur F, Wagner F, Welz A, Uberfuhr P, Briegel H, Reichart B. First experience with FK 506 for treatment of chronic pulmonary rejection. Transplant Proc. 1995 Jun;27(3):2009. No abstract available. PMID 7540775
- [Background] Kesten S, Chaparro C, Scavuzzo M, Gutierrez C. Tacrolimus as rescue therapy for bronchiolitis obliterans syndrome. J Heart Lung Transplant. 1997 Sep;16(9):905-12. PMID 9322139
- [Background] Speich R, Boehler A, Thurnheer R, Weder W. Salvage therapy with mycophenolate mofetil for lung transplant bronchiolitis obliterans: importance of dosage. Transplantation. 1997 Aug 15;64(3):533-5. doi: 10.1097/00007890-199708150-00027. PMID 9275125
- [Background] Whyte RI, Rossi SJ, Mulligan MS, Florn R, Baker L, Gupta S, Martinez FJ, Lynch JP 3rd. Mycophenolate mofetil for obliterative bronchiolitis syndrome after lung transplantation. Ann Thorac Surg. 1997 Oct;64(4):945-8. doi: 10.1016/s0003-4975(97)00845-x. PMID 9354506
- [Background] Diamond DA, Michalski JM, Lynch JP, Trulock EP 3rd. Efficacy of total lymphoid irradiation for chronic allograft rejection following bilateral lung transplantation. Int J Radiat Oncol Biol Phys. 1998 Jul 1;41(4):795-800. doi: 10.1016/s0360-3016(98)00113-8. PMID 9652840
- [Background] Higenbottam T, Jackson M, Woolman P, Lowry R, Wallwork J. The cough response to ultrasonically nebulized distilled water in heart-lung transplantation patients. Am Rev Respir Dis. 1989 Jul;140(1):58-61. doi: 10.1164/ajrccm/140.1.58. PMID 2502056
- [Background] Rivero DH, Lorenzi-Filho G, Pazetti R, Jatene FB, Saldiva PH. Effects of bronchial transection and reanastomosis on mucociliary system. Chest. 2001 May;119(5):1510-5. doi: 10.1378/chest.119.5.1510. PMID 11348961
- [Background] Tomkiewicz RP, App EM, Shennib H, Ramirez O, Nguyen D, King M. Airway mucus and epithelial function in a canine model of single lung autotransplantation. Chest. 1995 Jan;107(1):261-5. doi: 10.1378/chest.107.1.261. PMID 7813288
- [Background] Veale D, Glasper PN, Gascoigne A, Dark JH, Gibson GJ, Corris PA. Ciliary beat frequency in transplanted lungs. Thorax. 1993 Jun;48(6):629-31. doi: 10.1136/thx.48.6.629. PMID 8346493
- [Background] Herve P, Silbert D, Cerrina J, Simonneau G, Dartevelle P. Impairment of bronchial mucociliary clearance in long-term survivors of heart/lung and double-lung transplantation. The Paris-Sud Lung Transplant Group. Chest. 1993 Jan;103(1):59-63. doi: 10.1378/chest.103.1.59. PMID 8380268
- [Background] Blondeau K, Mertens V, Vanaudenaerde BA, Verleden GM, Van Raemdonck DE, Sifrim D, Dupont LJ. Nocturnal weakly acidic reflux promotes aspiration of bile acids in lung transplant recipients. J Heart Lung Transplant. 2009 Feb;28(2):141-8. doi: 10.1016/j.healun.2008.11.906. PMID 19201339
- [Background] Sweet MP, Herbella FA, Leard L, Hoopes C, Golden J, Hays S, Patti MG. The prevalence of distal and proximal gastroesophageal reflux in patients awaiting lung transplantation. Ann Surg. 2006 Oct;244(4):491-7. doi: 10.1097/01.sla.0000237757.49687.03. PMID 16998357
- [Background] Savarino E, Bazzica M, Zentilin P, Pohl D, Parodi A, Cittadini G, Negrini S, Indiveri F, Tutuian R, Savarino V, Ghio M. Gastroesophageal reflux and pulmonary fibrosis in scleroderma: a study using pH-impedance monitoring. Am J Respir Crit Care Med. 2009 Mar 1;179(5):408-13. doi: 10.1164/rccm.200808-1359OC. Epub 2008 Dec 18. PMID 19096004
- [Background] Sweet MP, Patti MG, Hoopes C, Hays SR, Golden JA. Gastro-oesophageal reflux and aspiration in patients with advanced lung disease. Thorax. 2009 Feb;64(2):167-73. doi: 10.1136/thx.2007.082719. PMID 19176842
- [Background] Benden C, Aurora P, Curry J, Whitmore P, Priestley L, Elliott MJ. High prevalence of gastroesophageal reflux in children after lung transplantation. Pediatr Pulmonol. 2005 Jul;40(1):68-71. doi: 10.1002/ppul.20234. PMID 15880421
- [Background] Palmer SM, Miralles AP, Howell DN, Brazer SR, Tapson VF, Davis RD. Gastroesophageal reflux as a reversible cause of allograft dysfunction after lung transplantation. Chest. 2000 Oct;118(4):1214-7. doi: 10.1378/chest.118.4.1214. PMID 11035701
- [Background] Rinaldi M, Martinelli L, Volpato G, Pederzolli C, Silvestri M, Pederzolli N, Arbustini E, Vigano M. Gastro-esophageal reflux as cause of obliterative bronchiolitis: a case report. Transplant Proc. 1995 Jun;27(3):2006-7. No abstract available. PMID 7792868
- [Background] Young LR, Hadjiliadis D, Davis RD, Palmer SM. Lung transplantation exacerbates gastroesophageal reflux disease. Chest. 2003 Nov;124(5):1689-93. doi: 10.1378/chest.124.5.1689. PMID 14605036
- [Background] Stovold R, Forrest IA, Corris PA, Murphy DM, Smith JA, Decalmer S, Johnson GE, Dark JH, Pearson JP, Ward C. Pepsin, a biomarker of gastric aspiration in lung allografts: a putative association with rejection. Am J Respir Crit Care Med. 2007 Jun 15;175(12):1298-303. doi: 10.1164/rccm.200610-1485OC. Epub 2007 Apr 5. PMID 17413126
- [Background] Meltzer AJ, Weiss MJ, Veillette GR, Sahara H, Ng CY, Cochrane ME, Houser SL, Sachs DH, Rosengard BR, Madsen JC, Wain JC, Allan JS. Repetitive gastric aspiration leads to augmented indirect allorecognition after lung transplantation in miniature swine. Transplantation. 2008 Dec 27;86(12):1824-9. doi: 10.1097/TP.0b013e318190afe6. PMID 19104429
- [Background] Hartwig MG, Appel JZ, Li B, Hsieh CC, Yoon YH, Lin SS, Irish W, Parker W, Davis RD. Chronic aspiration of gastric fluid accelerates pulmonary allograft dysfunction in a rat model of lung transplantation. J Thorac Cardiovasc Surg. 2006 Jan;131(1):209-17. doi: 10.1016/j.jtcvs.2005.06.054. Epub 2005 Dec 9. PMID 16399314
- [Background] Downing TE, Sporn TA, Bollinger RR, Davis RD, Parker W, Lin SS. Pulmonary histopathology in an experimental model of chronic aspiration is independent of acidity. Exp Biol Med (Maywood). 2008 Oct;233(10):1202-12. doi: 10.3181/0801-RM-17. Epub 2008 Jul 18. PMID 18641054
- [Background] Li B, Hartwig MG, Appel JZ, Bush EL, Balsara KR, Holzknecht ZE, Collins BH, Howell DN, Parker W, Lin SS, Davis RD. Chronic aspiration of gastric fluid induces the development of obliterative bronchiolitis in rat lung transplants. Am J Transplant. 2008 Aug;8(8):1614-21. doi: 10.1111/j.1600-6143.2008.02298.x. Epub 2008 Jun 28. PMID 18557728
- [Background] Hadjiliadis D, Davis RD, Lawrence CM, Rea JB, Tapson V, Brazer SR, Palmer SM. Associatioin of Bronchiolitis Obliterans Syndrome (BOS) With Gastroesophageal Reflux Disease (GERD) in Lung Transplant Recipients. Am J Respir Crit Care Med. 2001;163(5):A325.
- [Background] Hadjiliadis D, Duane Davis R, Steele MP, Messier RH, Lau CL, Eubanks SS, Palmer SM. Gastroesophageal reflux disease in lung transplant recipients. Clin Transplant. 2003 Aug;17(4):363-8. doi: 10.1034/j.1399-0012.2003.00060.x. PMID 12868994
- [Background] Cantu E 3rd, Appel JZ 3rd, Hartwig MG, Woreta H, Green C, Messier R, Palmer SM, Davis RD Jr. J. Maxwell Chamberlain Memorial Paper. Early fundoplication prevents chronic allograft dysfunction in patients with gastroesophageal reflux disease. Ann Thorac Surg. 2004 Oct;78(4):1142-51; discussion 1142-51. doi: 10.1016/j.athoracsur.2004.04.044. PMID 15464462
- [Background] D'Ovidio F, Mura M, Tsang M, Waddell TK, Hutcheon MA, Singer LG, Hadjiliadis D, Chaparro C, Gutierrez C, Pierre A, Darling G, Liu M, Keshavjee S. Bile acid aspiration and the development of bronchiolitis obliterans after lung transplantation. J Thorac Cardiovasc Surg. 2005 May;129(5):1144-52. doi: 10.1016/j.jtcvs.2004.10.035. PMID 15867792
- [Background] S.C Murthy1 ERN, D.P. Mason1, M.M. Budev2, A.I. Nunez1, L. Thuita3, J.T. Chapman2, G.B. Pettersson1, E.H. Blackstone1, 3 Preoperative Gastroesophageal Reflux Impacts Early Outcomes after Lung Transplantation. The Journal of Heart and Lung Transplantation. 2009 February 28(2):S214.
- [Background] Lau CL, Palmer SM, Hadjiliadis D, Pappas TN, Eubanks W, Davis RD. Anti-reflux surgery improves pulmonary function in lung transplant recipients. J Heart Lung Transplant. 2002;21(1):108.
- [Background] Davis RD Jr, Lau CL, Eubanks S, Messier RH, Hadjiliadis D, Steele MP, Palmer SM. Improved lung allograft function after fundoplication in patients with gastroesophageal reflux disease undergoing lung transplantation. J Thorac Cardiovasc Surg. 2003 Mar;125(3):533-42. doi: 10.1067/mtc.2003.166. PMID 12658195
- [Background] Hartwig MG, Appel JZ, Davis RD. Antireflux surgery in the setting of lung transplantation: strategies for treating gastroesophageal reflux disease in a high-risk population. Thorac Surg Clin. 2005 Aug;15(3):417-27. doi: 10.1016/j.thorsurg.2005.03.001. PMID 16104132